CLINICAL TRIAL: NCT02637713
Title: Radiofrequency Energy Delivery to the Lower Esophageal Sphincter (Stretta) in Sleeve Gastrectomy Patients With GERD
Brief Title: Management of Reflux After Sleeve Using Stretta
Acronym: MaRSS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Accrual
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-5661a
Record Dates: First submitted 2015-11-16; First posted 2015-12-22 (Estimated); Results first posted 2023-05-08 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-12

CONDITIONS: GERD; Morbid Obesity
Keywords: GERD; sleeve gastrectomy; reflux; morbidly obese
MeSH Terms: conditions — Gastroesophageal Reflux; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Radiofrequency Energy to the Lower Esophageal Sphincter (LES) (Experimental): All patients that have undergone sleeve gastrectomy as treatment for obesity that have developed severe reflux symptoms will be treated with Stretta (FDA approved device for the management of GERD) and evaluated prospectively for resolution/improvement of reflux symptoms.
  Interventions: Device: Stretta; Procedure: Radiofrequency (RF) Energy to the LES (Stretta Procedure)

INTERVENTIONS:
Device: Stretta — Stretta is an FDA approved device that delivers Radiofrequency energy delivery to the lower esophageal sphincter. It is approved for the management of GRED.
Procedure: Radiofrequency (RF) Energy to the LES (Stretta Procedure) — The Stretta procedure is performed endoscopically under moderate sedation or general anesthesia which uses radiofrequency (RF) energy applied to the lower esophagus over 14 minutes per FDA approved procedures.

SUMMARY:
Gastroesophageal reflux disease (GERD) is a frequently seen entity after sleeve gastrectomy. Management of GERD after sleeve is difficult given limited treatment modalities. Stretta is an endoscopic FDA approved device that improves symptoms of GERD, there is minimal information about its use on patients after sleeve. This registry will attempt to get information regarding the treatment of reflux using Stretta after sleeve gastrectomy.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is a widely prevalent medical disorder in the United States with a spectrum of treatment options ranging from dietary modification, to various pharmacologic treatments, to an array of available surgical and endoscopic procedures. There is a well-described correlation between obesity and symptoms of GERD. The morbidly obese patients undergoing evaluation for bariatric surgery are to characterize any GERD-like symptoms as this will assist in directing surgical therapy. Generally, it is recommended that patients with severe GERD undergo Roux-en-Y gastric bypass(RYGB) rather than a sleeve gastrectomy (SG) as RYGB has proven to be the most effective surgical treatment for GERD in the morbidly obese patient. The number of bariatric procedures performed in the United States has increased significantly in the recent years. Out of all bariatric procedures SG is the most commonly performed in the United States, as it has proven to be a very safe procedure with excellent weight loss. However, the incidence of de novo GERD and the effect of SG on patients with preexisting GERD remain controversial. Although some authors report high incidence of de novo GERD and worsening of previous reflux symptoms, there is also data showing improvement of symptoms post SG. Management of GERD after SG poses an interesting challenge, as traditional invasive procedures like Nissen fundoplication are not available due to an altered gastric anatomy. The alternative is to perform a conversion to RYGB, which represents increased morbidity to patient and significant cost.

A large number of endoscopic procedures have been introduced in the past for the management of GERD as an alternative to the surgical anti-reflux procedures with various degrees of success. One of the few non-invasive methods for managing GERD that is still available on the market and widely used is Stretta. Stretta delivers Radio Frequency energy (RFe) to the LES resulting in increased LES pressure. In 2000, the FDA approved the Stretta system for treatment of GERD. Stretta allows an alternative for treatment in patients who are not willing or able to undergo surgery. The Society of American Gastrointestinal and Endoscopic Surgeons (SAGES) published clinical practice guidelines that endorsed Stretta as an appropriate therapy for treatment of GERD in patients >18, with at least 6 months of symptoms partially or completely responsive to pharmacotherapy and who are unable or unwilling to undergo laparoscopic Nissen fundoplication. There are to date no studies evaluating the use of Stretta in management of patients with GERD symptoms after sleeve gastrectomy.

The investigators will study sleeve gastrectomy patients with GERD symptoms and if considered candidates for Stretta all patients will be enrolled in data collection cohort and followed prospectively with symptom questionnaire and quality of life scores for improvement of symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic reflux: (heartburn, chest discomfort, asthma/chronic cough, laryngitis, nocturnal aspiration or regurgitation)
2. On a PPI with GERD-related symptoms
3. On a PPI but like to discontinue them

Exclusion Criteria:

1. Age <18 or > 80
2. History of a severe psychiatric disorder: including suicidal ideation, or admission to a psychiatric institution.
3. Unable or unwilling to consent for an invasive procedure.
4. History of intestinal leak after surgery.
5. History of revisional bariatric surgery
6. Significant sleeve abnormalities such and twist or large fundus
7. Hiatal hernia(>2cm)
8. Pregnancy
9. Inability to comply with study protocols and procedures
10. Esophageal stricture, Eosinophilic Esophagitis or Achalasia
11. Prior esophageal surgery or therapy for Barrett's Esophagus
12. Grades 3 or 4 esophagitis
13. Gastric or esophageal varices
14. History of obstruction of the small bowel or inflammatory bowel disease
15. Pacemaker or implanted cardiac defibrillator
16. Coagulopathy or use of anticoagulants
17. ASA classification >3
18. Scleroderma or other connective diseases
19. Use of immunosuppressive medications.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Moran-Atkin, MD, Principal Investigator — Assistant Professor
Locations (13):
- United States (13):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - Norwalk Hospital, Norwalk, Connecticut
  - Gastroenterology Clinic of Acadiana, Lafayette, Louisiana
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Health System, Durham, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic Health System, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann-Texas Medical Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiofrequency Energy to the Lower Esophageal Sphincter (LES)
Started | 5
Completed | 3
Not Completed | 2
Not completed — Screen Failure | 2

BASELINE CHARACTERISTICS:
Arm/Group | Radiofrequency Energy to the Lower Esophageal Sphincter (LES)
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Black or African-American | 1
  White Non-Hispanic | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Improved Symptoms Based on Reflux Symptom Index (RSI) Score
Description: RSI scores will be used to determine whether patients achieved at least a 50% reduction in symptoms as compared to baseline. Patients will be provided a 9-item questionnaire and asked to rate the score that best applies to their symptoms on a 6 point scale ranging from 0 = No Problem to 5 = Severe Problem.
Time Frame: 6 months
Population: Study was terminated early and no 6 month RSI data were collected. As such, there were no RSI scores to aggregate and report.
Arm/Group | Radiofrequency Energy to the Lower Esophageal Sphincter (LES)
Number analyzed (Participants) | 0

2. Primary Outcome: Number of Patients With Improved Symptoms Based on Reflux Severity Index (RSI) Score
Description: as for outcome 1
Time Frame: 12 months
Population: Study was terminated early and no 12 month RSI data were collected. As such, there were no RSI scores to aggregate and report.
Arm/Group | Radiofrequency Energy to the Lower Esophageal Sphincter (LES)
Number analyzed (Participants) | 0

3. Primary Outcome: Number of Patients With Improved Symptoms Based on Reflux Severity Index (RSI) Score
Description: as for outcome 1
Time Frame: 24 months
Population: Study was terminated early and no 24 month RSI data were collected. As such, there were no RSI scores to aggregate and report.
Arm/Group | Radiofrequency Energy to the Lower Esophageal Sphincter (LES)
Number analyzed (Participants) | 0

4. Primary Outcome: Number of Patients With Improved Symptoms Based on GERD Health Related Quality of Life (GERD-HRQL) Questionnaire Score
Description: GERD-HRQL scores will be used to determine whether patients achieved at least a 50% reduction in symptoms as compared to baseline. Patients will be provided a 15-item questionnaire and asked to rate the score that best applies to their symptoms on a 6 point scale ranging from 0 to 5 (overall range from 0-75) with higher scores indicative of worsening symptoms.
Time Frame: 6 months
Population: Study was terminated early and no 6 month GERD-HRQL data were collected. As such, there were no results to aggregate and report.
Arm/Group | Radiofrequency Energy to the Lower Esophageal Sphincter (LES)
Number analyzed (Participants) | 0

5. Primary Outcome: Number of Patients With Improved Symptoms Based on GERD Health Related Quality of Life (GERD-HRQL) Questionnaire Score
Description: as for outcome 4
Time Frame: 12 months
Population: Study was terminated early and no 12 month GERD-HRQL data were collected. As such, there were no results to aggregate and report.
Arm/Group | Radiofrequency Energy to the Lower Esophageal Sphincter (LES)
Number analyzed (Participants) | 0

6. Primary Outcome: Number of Patients With Improved Symptoms Based on GERD Health Related Quality of Life (GERD-HRQL) Questionnaire Score
Description: as for outcome 4
Time Frame: 24 months
Population: Study was terminated early and no 24 month GERD-HRQL data were collected. As such, there were no results to aggregate and report.
Arm/Group | Radiofrequency Energy to the Lower Esophageal Sphincter (LES)
Number analyzed (Participants) | 0

7. Secondary Outcome: Esophageal pH Levels
Description: All patients will have pH monitoring conducted at baseline pre-procedurally. The number of patients with abnormal pH levels will be tabulated. Bravo capsule monitoring will be used for evaluation.
Time Frame: Baseline
Population: Esophageal samples were not collected and therefore there was no esophageal pH results to report.
Arm/Group | Radiofrequency Energy to the Lower Esophageal Sphincter (LES)
Number analyzed (Participants) | 0

8. Secondary Outcome: Esophageal pH Levels
Description: If esophageal pH levels at baseline are determined to have been abnormal, the number of patients with symptomatic GERD demonstrating an improvement in esophageal pH exposure following sleeve gastrectomy will be assessed. Bravo capsule monitoring will be used for evaluation.
Time Frame: 6 months
Population: Study was terminated early. Esophageal samples were not collected and therefore there was no esophageal pH results to report.
Arm/Group | Radiofrequency Energy to the Lower Esophageal Sphincter (LES)
Number analyzed (Participants) | 0

9. Secondary Outcome: Esophageal pH Levels
Description: as for outcome 8
Time Frame: 12 months
Population: as for outcome 8
Arm/Group | Radiofrequency Energy to the Lower Esophageal Sphincter (LES)
Number analyzed (Participants) | 0

10. Secondary Outcome: Use of Anti-reflux Medication
Description: The number of patients using anti-reflux medications will be tabulated.
Time Frame: Baseline
Population: Study was terminated early and data related to the use of anti-reflux medications was not collected. As such, there were no related anti-reflux medication data to aggregate and report.
Arm/Group | Radiofrequency Energy to the Lower Esophageal Sphincter (LES)
Number analyzed (Participants) | 0

11. Secondary Outcome: Cessation or Decreased Use of Anti-reflux Medication
Description: The number of patients who demonstrate a complete cessation or decrease in use of anti-reflux medications will be tabulated.
Time Frame: 6 months
Population: Study was terminated early and data related to the cessation or decreased use of anti-reflux medications was not collected. As such, there were no related anti-reflux medication data to aggregate and report.
Arm/Group | Radiofrequency Energy to the Lower Esophageal Sphincter (LES)
Number analyzed (Participants) | 0

12. Secondary Outcome: Gastric Emptying Study
Description: A Gastric emptying study will be conducted for all patients at 1, 2, 3, and 4 hours. Patients with severe gastroparesis (>50% retention at 4 hours) will be excluded from study
Time Frame: Baseline (up to 4 hours)
Population: Study was terminated early and the gastric emptying study was not collected. As such, there were no related gastric emptying data to aggregate and report.
Arm/Group | Radiofrequency Energy to the Lower Esophageal Sphincter (LES)
Number analyzed (Participants) | 0

13. Secondary Outcome: Determination of Gastric Dysmotility as a Contributory Factor in GERD Following Sleeve Gastrectomy
Description: If gastric dysmotility is determined to have been abnormal at baseline, the gastric emptying study will be repeated at 6 months to evaluate Gastric Dysmotility will be evaluated as a contributory factor in GERD following sleeve gastrectomy.
Time Frame: 6 months
Population: Study was terminated early and data related to gastric dysmotility as a contributing factor to GERD was not collected. As such, there were no 6 month gastric dysmotility results to aggregate and report.
Arm/Group | Radiofrequency Energy to the Lower Esophageal Sphincter (LES)
Number analyzed (Participants) | 0

14. Secondary Outcome: Determination of Gastric Dysmotility as a Contributory Factor in GERD Following Sleeve Gastrectomy
Description: If gastric dysmotility is determined to have been abnormal at baseline, the gastric emptying study will be repeated at 12 months to evaluate Gastric Dysmotility will be evaluated as a contributory factor in GERD following sleeve gastrectomy.
Time Frame: 12 months
Population: Study was terminated early and data related to gastric dysmotility as a contributing factor to GERD was not collected. As such, there were no 12 month gastric dysmotility results to aggregate and report.
Arm/Group | Radiofrequency Energy to the Lower Esophageal Sphincter (LES)
Number analyzed (Participants) | 0

15. Secondary Outcome: EGD Abnormalities
Description: An EGD will be obtained for all patients at baseline. Biopsies of any suspicious lesions and any evidence of esophagitis will be obtained and scored in accordance with Los Angeles classification as either Grade A, Grade B, Grade C, or Grade D lesions with each grade denoting progressively more severe pathophysiology.
Time Frame: Baseline
Population: Biopsies were not obtained at baseline and, as such, there were no corresponding results to analyze and report.
Arm/Group | Radiofrequency Energy to the Lower Esophageal Sphincter (LES)
Number analyzed (Participants) | 0

16. Secondary Outcome: EGD Abnormalities
Description: In those patients identified to have abnormal esophageal pathology at baseline, biopsies of any suspicious lesions and any evidence of esophagitis will be obtained and scored in accordance with Los Angeles classification as either Grade A, Grade B, Grade C, or Grade D lesions with each grade denoting progressively more severe pathology. The number of patients demonstrating objective histologic improvement or resolution of esophagitis will be determined.
Time Frame: 6 months
Population: Study was terminated early. Biopsies were not obtained at 6 months and, as such, there were no corresponding results to analyze and report.
Arm/Group | Radiofrequency Energy to the Lower Esophageal Sphincter (LES)
Number analyzed (Participants) | 0

17. Secondary Outcome: EGD Abnormalities
Description: as for outcome 16
Time Frame: 12 months
Population: Study was terminated early. Biopsies were not obtained at 12 months and, as such, there were no corresponding results to analyze and report.
Arm/Group | Radiofrequency Energy to the Lower Esophageal Sphincter (LES)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Following Stretta procedure through week 4 and every 3 months thereafter up to 24 months
Arm/Group | Radiofrequency Energy to the Lower Esophageal Sphincter (LES)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT02637713/Prot_SAP_000.pdf